CLINICAL TRIAL: NCT05511376
Title: Comparison of Diet, Exercise, and Auricular Vagus Nerve Stimulation Efficacy for Weight Reduction in Obese Individuals
Brief Title: Comparison of Different Weight Loss Methods in Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Gozde In, EXPERT PHYSIOTHERAPIST AND DIETICIAN, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAUGOZDEIN1318303
Record Dates: First submitted 2022-08-04; First posted 2022-08-23 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DIET (Active Comparator): Personal nutrition programs were prepared according to ideal body weight, with protein intake as 30% of total daily calories or 1-1.2 g/kg.
  Interventions: Behavioral: DIET
- EXERCISE (Active Comparator): A pre-exercise breathing exercise study was planned.
  Exercise:
  It was planned to apply the Moderate Resistant Exercise Protocol (3 days a week for 60 minutes) and as aerobic exercise, walking 5 days a week (150 minutes / week) as 30 minutes / day.
  Interventions: Behavioral: EXERCISE
- AURICULAR VAGUS NERVE STIMULATION (Active Comparator): The Vagustim device was applied in Biphasic, Frequency 10 Hz, Modulation mode, with a pulse width of 300 μs, for 30 minutes /3 days/week by keeping the current intensity constant where the participants felt comfortable.
  It will be applied as bilateral VSS from the tragus and turbinate parts of the ear.
  Interventions: Device: AURICULAR VAGUS NERVE STIMULATION

INTERVENTIONS:
Device: AURICULAR VAGUS NERVE STIMULATION — For 4 weeks With the Vagustim device, in Biphasic, Frequency 10 Hz, Modulation mode, the pulse width of 300 μs, where the participants feel comfortable, the current intensity is kept constant for 30 minutes / 3 days/week. It will be applied as bilateral VSS from the tragus and turbinate parts of the ear.
  Other Names: Vagustim
  Arms: AURICULAR VAGUS NERVE STIMULATION
Behavioral: DIET — For 4 weeks, Protein intake to 30% of total daily calories or 1-1.2 g/kg Personal nutrition program created for ideal body weight (by BMI values for age)
  Other Names: A Mediterranean-style, protein-based diet program
  Arms: DIET
Behavioral: EXERCISE — Exercise: Moderate Resistance Exercise Protocol (60 min 3 days a week )+ 30 min/day as aerobic exercise ( 5 days a week)
  Other Names: Moderate Resistance Exercise and Aerobic Exercise
  Arms: EXERCISE

SUMMARY:
Although obesity is a rapidly increasing epidemic worldwide, it is associated with many health-related comorbidities. As a result of the developments in social life and observes the sedentary life in individuals, an effect of the age of technology the fact that this epidemic will cause even massive health problems in the coming period affecting the health systems of countries and indirectly their economies that, This situation necessitates the creation of alternative treatment methods for the prevention of obesity. This study aims to determine the effect of a therapy approach that can be applied to the vagus nervous system, which is associated with many organs and systems, on weight loss and general health. As an alternative treatment against lifestyle changes such as diet and exercise, individuals have made for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 - 65
* Being in the stage I, II and III obesity class

Exclusion Criteria:

* Those with unstable DM
* Those with stage II hypertension
* Those who have had cardiovascular disease (especially those who have had an attack)
* Those with pulmonary disease
* Those with kidney disease
* Orthopedic restrictions
* Those with MND
* Those tied to the chair

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-26 (Estimated)

PRIMARY OUTCOMES:
Body Analysis | Study start
  BIA measurements include (BMI (kg/m2)).
Body Analysis | 2nd week
  BIA measurements include (BMI (kg/m2)).
Body Analysis | 4th week
  BIA measurements include (BMI (kg/m2)).
Body Analysis | Study start
  BIA measurements include (Weight ( kg), Muscle and fat mass (kg), Body bone and fluid mass (kg), such as).
Body Analysis | 2nd week
  BIA measurements include (Weight ( kg), Muscle and fat mass (kg), Body bone and fluid mass (kg), such as).
Body Analysis | 4th week
  BIA measurements include (Weight ( kg), Muscle and fat mass (kg), Body bone and fluid mass (kg), such as).
Body Analysis | Study start
  BIA measurements include (Muscle and fat percentage (%) such as).
Body Analysis | 2nd week
  BIA measurements include (Muscle and fat percentage (%) such as).
Body Analysis | 4th week
  BIA measurements include (Muscle and fat percentage (%) such as).
Body Analysis | Study start
  BIA measurement include (Body density (mg/dl)).
Body Analysis | 2nd week
  BIA measurement include (Body density (mg/dl)).
Body Analysis | 4th week
  BIA measurement include (Body density (mg/dl)).
Body Analysis | Study start
  BIA measurement include (internal adiposity).
Body Analysis | 2nd week
  BIA measurement include (internal adiposity).
Body Analysis | 4th week
  BIA measurement include (internal adiposity).
Anthropometric Measurements | Study start
  It includes length (m) measurement.
Anthropometric Measurements | 2nd week
  It includes length (m) measurement.
Anthropometric Measurements | 4th week
  It includes length (m) measurement.
Anthropometric Measurements | Study start
  It includes waist (cm), hip (cm), upper arm (cm), thigh circumference (cm) and Skinfold thickness(cm) measurements.
Anthropometric Measurements | 2nd week
  It includes waist (cm), hip (cm), upper arm (cm), thigh circumference (cm) and Skinfold thickness(cm) measurements.
Anthropometric Measurements | 4th week
  It includes waist (cm), hip (cm), upper arm (cm), thigh circumference (cm) and Skinfold thickness(cm) measurements.
Anthropometric Measurements | Study start
  It includes waist-hip ratio measurements.
Anthropometric Measurements | 2nd week
  It includes waist-hip ratio measurements.
Anthropometric Measurements | 4th week
  It includes waist-hip ratio measurements.
Biochemical parameters | Study start & 4th week
  It includes fasting blood sugar (mg/dL) value.
Biochemical parameters | Study start
  It includes fasting blood sugar (mg/dL) value.
Biochemical parameters | 4th week
  It includes HDL (mg/dL), LDL (mg/dL), TG (mg/dL), and Total cholesterol (mg/dL) values.
Biophysical Methods | Study start
  It includes 5 X Sit-to-Stand Up test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 2nd week
  It includes 5 X Sit-to-Stand Up test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 4th week
  It includes 5 X Sit-to-Stand Up test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | Study start
  It includes the Stair Climb test (sec). ( It shows the temporal variation values in performing a particular activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 2nd week
  It includes the Stair Climb test (sec). ( It shows the temporal variation values in performing a particular activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 4th week
  It includes the Stair Climb test (sec). ( It shows the temporal variation values in performing a particular activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | Study start
  It includes The Timed Up and Go Test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 2nd week
  It includes The Timed Up and Go Test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
Biophysical Methods | 4th week
  It includes The Timed Up and Go Test (sec). ( It show the temporal variation values in performing a certain activity. Functional activity and used to assess balance. Completion of test activity in a short time indicates positive development.)
6-Min Walk Test | Study start
  The 6-minute walk test includes value walking distance (m). (Increased walking distance indicates that functional values develop positively.)
6-Min Walk Test | 2nd week
  The 6-minute walk test includes value walking distance (m). (Increased walking distance indicates that functional values develop positively.)
6-Min Walk Test | 4th week
  The 6-minute walk test includes value walking distance (m). (Increased walking distance indicates that functional values develop positively.)
6-Min Walk Test | Study start
  The 6-minute walk test includes value Blood pressure (mmHg) measurements. (High blood pressure measurements approaching the normal value indicate that functional values develop positively.)
6-Min Walk Test | 2nd week
  The 6-minute walk test includes value Blood pressure (mmHg) measurements. (High blood pressure measurements approaching the normal value indicate that functional values develop positively.)
6-Min Walk Test | 4th week
  The 6-minute walk test includes value Blood pressure (mmHg) measurements. (High blood pressure measurements approaching the normal value indicate that functional values develop positively.)
6-Min Walk Test | Study start
  The 6-minute walk test includes value Modified Borg Dyspnea and Fatigue Scores. (Decreased dyspnea and fatigue scores indicate that functional values develop positively.)
6-Min Walk Test | 2nd week
  The 6-minute walk test includes value Modified Borg Dyspnea and Fatigue Scores. (Decreased dyspnea and fatigue scores indicate that functional values develop positively.)
6-Min Walk Test | 4th week
  The 6-minute walk test includes value Modified Borg Dyspnea and Fatigue Scores. (Decreased dyspnea and fatigue scores indicate that functional values develop positively.)
6-Min Walk Test | Study start
  The 6-minute walk test includes value Heart Rate. (Heart rate values being within the normal range for age indicate that functional values develop positively.)
6-Min Walk Test | 2nd week
  The 6-minute walk test includes value Heart Rate. (Heart rate values being within the normal range for age indicate that functional values develop positively.)
6-Min Walk Test | 4th week
  The 6-minute walk test includes value Heart Rate. (Heart rate values being within the normal range for age indicate that functional values develop positively.)
6-Min Walk Test | Study start
  The 6-minute walk test includes value O2 saturation (mmHg). (Increased O2 saturation indicates that functional values develop positively.)
6-Min Walk Test | 2nd week
  The 6-minute walk test includes value O2 saturation (mmHg). (Increased O2 saturation indicates that functional values develop positively.)
6-Min Walk Test | 4th week
  The 6-minute walk test includes value O2 saturation (mmHg). (Increased O2 saturation indicates that functional values develop positively.)
Handgrip strength test | Study start
  The Handgrip strength test (kg) measurement evaluates muscle strength.
Handgrip strength test | 2nd week
  The Handgrip strength test (kg) measurement evaluates muscle strength.
Handgrip strength test | 4th week
  The Handgrip strength test (kg) measurement evaluates muscle strength.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (Short Form- IPAQ) | Study start, 2nd & 4th week
  It has been used to examine physical activity levels. (Weekly physical activity levels are measured by MET value calculations. An increase in MET values indicates an increase in activity.)
Quality of Life Questionnaire (Short Form - SF-36) | Study start, 2nd & 4th week
  It was used to evaluate the effect of weight on quality of life. (It is evaluated in the range of 0 - 100 points. Energy/vitality, physical function, mental health, general health perception, social functionality scores show a positive development as they approach the maximum value. Physical role difficulty, emotional role difficulty and Pain scores show a positive development as they approach the minimum value.)
Food Cravings Questionnaire (FCQ) | Study start & 4th week
  It was used to determine the cravings for foods. (In the scale, a scoring system between 39-234 points is used for sub-dimensions.It shows that there is a positive development as the scale approaches the minimum result.)
Visual Analog Scale (VAS) | Study start, 2nd & 4th week
  It was used to determine the cravings for foods. (A scoring system from 0 to 10 is used.It shows that there is a positive development as the scale approaches the minimum result.)

CONTACTS AND LOCATIONS:
Overall Officials: Gözde IN, Principal Investigator — Bahçeşehir University
Locations (1):
- Avicenna Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No